CLINICAL TRIAL: NCT02113553
Title: ANTI-MULLERIAN HORMONE (AMH) AS A MARKER OF OVARIAN RESERVE IN YOUNG BREAST CANCER PATIENTS RECEIVING CHEMOTHERAPY + GnRH ANALOGUE
Brief Title: Anti-Mullerian Hormone (AMH) as Marker of Ovarian Reserve
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: target population not reached
Sponsor: Armando Santoro, MD (Other)
Responsible Party: Sponsor-Investigator, Armando Santoro, MD, Principal Investigator, Istituto Clinico Humanitas
Organization: Istituto Clinico Humanitas (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ONC-2012-002
Record Dates: First submitted 2013-05-27; First posted 2014-04-14 (Estimated); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Triptorelin (Experimental): Triptorelin 3.75 administered every 28 days, for 4 to 7 injections depending on the number of cycles of chemotherapy
  Interventions: Drug: Triptorelin

INTERVENTIONS:
Drug: Triptorelin — Triptorelin administered once every 28 days in addition to chemotherapy
  Other Names: Decapeptyl; Gonapeptyl

SUMMARY:
This is a multicentre, prospective study willing to evaluate AMH levels changes in response to chemotherapy plus GnRHa.

In the present study we propose to determine AMH levels in breast cancer patients, aged <40yrs receiving adjuvant chemotherapy and ovarian suppression by means of GnRHa with the aim to assess the role of AMH as surrogate marker of the preservation of ovarian reserve exerted by GnRHa.

DETAILED DESCRIPTION:
Patients will receive 4 to 8 cycles of chemotherapy according to Institutional guidelines. Triptorelin 3.75 will be administered as an intramuscular injection before chemotherapy and every 28 days thereafter for all the duration of chemotherapy in patients with ER negative tumors and for 2 to 5 years in patients with ER positive tumors according to Institutional guidelines. Patients with ER+ve tumour will receive tamoxifen for 5 years at the end of chemotherapy as standard care. A blood sample will be drawn after signed informed consent to determine baseline AMH levels. A blood sample for determination of AMH levels will be collected at the end of chemotherapy and at 12 months after the end of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects, aged <40yr at the time of breast cancer diagnosis
2. Diagnosis of operable breast cancer any T and N, any ER
3. Patients candidate to adjuvant chemotherapy for 4-8 cycles.
4. Patients compliant to adhere to all protocol procedures.
5. Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 28 days prior to the start of the study treatment.
6. Negative pregnancy test at the study enrolment; fertile women must use effective contraception during chemotherapy
7. Patients must be able to understand and sign written informed consent.

   -

Exclusion Criteria:

1. Presence of distant metastasis
2. Clinically significant cardiovascular disease
3. Psychological or social conditions which might affect study compliance
4. Unstable neurologic function
5. Patients with known allergy to any of the components of the study medication
6. Pregnancy or lactation
7. Any condition that, in the opinion of the physician is likely to affect inclusion of the subject into the study.

Max Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2013-05; Primary Completion 2016-05 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
AMH in response to chemotherapy plus GnRHa | 18 months
  To evaluate AMH levels changes in response to chemotherapy plus GnRHa in order to assess the role of AMH as surrogate marker of the preservation of ovarian reserve exerted by GnRHa

SECONDARY OUTCOMES:
AMH and menstrual cycle | 18 months
  To correlate AMH behaviour with recovery of menstrual cycle (in the ER negative cohort);
AMH after chemotherapy | 18 months
  To compare AMH levels obtained at the end of chemotherapy and at 12 months after the end of chemotherapy in the two cohorts of ER positive and ER negative patients
AMH levels >0.2 ng/mL at the 12-month time point | 18 months
  Evaluate the proportion of patients with AMH levels >0.2 ng/mL at the 12-month time point.

CONTACTS AND LOCATIONS:
Overall Officials: Armando Santoro, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milan, Italy